CLINICAL TRIAL: NCT05859763
Title: 99mTc-Labeled FAPI SPECT Imaging in Pulmonary Fibrosis
Brief Title: 99mTc-HFAPI SPECT/CT in Pulmonary Fibrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TcHFAPIPF
Record Dates: First submitted 2023-05-05; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients diagnosed with pulmonary fibrosis (Experimental): Patients of Pulmonary Fibrosis SPECT/CT imaging: The patients were subcutaneously injected with 99mTc-HFAPI and underwent SPECT/CT imaging.
  Interventions: Drug: 99mTc-HFAPI

INTERVENTIONS:
Drug: 99mTc-HFAPI — Each patient receive a intravenous injection of 99mTc-HFAPI, and undergo SPECT/CT scan within specified time.

SUMMARY:
This prospective study will investigate the potential usefulness of 99mTc labeled FAPI SPECT/CT in the diagnosis, treatment response assessment, and follow-up of pulmonary fibrosis.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis refers to a specific form of chronic fibrous interstitial pneumonia that occurs spontaneously, limited to the lung, and shows features of usual interstitial pneumonia on high resolution computed tomography and histological examination. Radionuclide labeled FAPI has been developed as a new tracer for tumor and inflammatory lesions imaging. Recent studies have shown that FAPI PET/CT imaging is a promising new imaging method for pulmonary fibrosis. HFAPI is obtained by conjugating 99mTc-chelator moiety (6-hydrazinonicotinamide, HYNIC) with FAP targeting moiety. The aim of this study is to investigate the location and extent of 99mTc labeled FAPI tracer (99mTc-HFAPI) in normal and fibrotic lung tissue of patients with pulmonary fibrosis, and to explore the clinical significance of 99mTc-HFAPI SPECT/CT in the diagnosis, treatment response evaluation and follow-up of pulmonary fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* suspected or confirmed pulmonary fibrosis patients;
* signed written consent.

Exclusion Criteria:

* pregnancy;
* breastfeeding;
* known allergy against FAPI
* any medical conditions that are considered by the investigator to be likely to seriously interfere with study compliance

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-12-12 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | through study completion, an average of 1.5 years
  Qualitative and semi-quantitative analysis (T/N ratio of lesions and adjacent normal tissue, and early and late imaging) of 99mTc-HFAPI SPECT/CT for pulmonary fibrosis

CONTACTS AND LOCATIONS:
Locations (1):
- Peking union medical college hospital, Beijing, Dongcheng, China